CLINICAL TRIAL: NCT03506282
Title: The Effects of Listening to Music During Running on Ground Contact Forces and Running Mechanics: the "IMPACT Factor" Trial
Brief Title: Does Listening to Music Alter the Running Mechanics?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Professor Franca Deriu, Associate Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: USassari
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Running biomechanics; Vertical loading rate; Music exercise; Gait analysis
MeSH Terms: interventions — Running

STUDY DESIGN:
Intervention Model Description: The experimental conditions to be tested in each subject will be: 0, running with no music; 1, running and listening to audio track resembling normal outdoor noise (70 dB); 2, running with music at moderate volume (80 dB); 3, running with music at moderate to high volume (85 dB). The experimental conditions will be carried out in random order, with a wash-out period of 10 minutes, to ensure the return to the auditory and vestibular baseline.
  Depending on the random sequence generated, the subject will undergo the four conditions in the specified order. Each condition will be completed with the three steps lasting 2 mins each (A, running at 6 km/h; B, running at 8 km/h; C, running at 10 km/h) and carried out at 1-min time interval in between, before proceeding to the next one. A complete rest of 10 minutes will be allowed among the conditions to restore the physiological state of the auditory and vestibular systems and to recover from the submaximal running effort.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants and the research assistant operator who will deliver the experimental conditions will not be masked to the condition whilst the outcome assessor, the statistician and the principal investigator will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No music (No Intervention): The participants will be required to run on a treadmill at 3 different speeds (6-8-10 km/h) with no music.
- Traffic audio track (Active Comparator): In addition to running on the treadmill, participants will be listening to an audio track resembling normal outdoor noise (70 dB) through earphones connected to a mobile phone.
  Interventions: Other: Running while listening to a traffic audio track
- Music at moderate volume (Experimental): In addition to running on the treadmill, participants will be listening to music at a moderate volume (80 dB) through earphones connected to a mobile phone.
  Interventions: Other: Running with music at moderate volume
- Music at moderate-to-high volume (Experimental): In addition to running on the treadmill, participants will be listening to music at a moderate-to-high volume (85 dB) through earphones connected to a mobile phone.
  Interventions: Other: Running with music at moderate-to-high volume

INTERVENTIONS:
Other: Running while listening to a traffic audio track — While running three 2-minute sets at different velocities (6, 8 and 10 km/h, respectively) on a sensorized treadmill, each participant will be exposed via earphones to an audio track resembling average outdoor conditions (70 dB).
  Other Names: Traffic audio track
  Arms: Traffic audio track
Other: Running with music at moderate volume — While running three 2-minute sets at different velocities (6, 8 and 10 km/h, respectively) on a sensorized treadmill, each participant will be provided the same music track ("We take care of our own", by Bruce Springsteen from the "Wrecking Ball" album, 2012). The music track will be given at a moderate volume (80 dB).
  Other Names: Music at moderate volume
  Arms: Music at moderate volume
Other: Running with music at moderate-to-high volume — While running three 2-minute sets at different velocities (6, 8 and 10 km/h, respectively) on a sensorized treadmill, each participant will be provided the same music track ("We take care of our own", by Bruce Springsteen from the "Wrecking Ball" album, 2012). The music track will be given at a moderate-to-high volume (85 dB).
  Other Names: Music at moderate-to-high volume
  Arms: Music at moderate-to-high volume

SUMMARY:
The purpose of this study is to determine whether in healthy subjects listening to music while running influences the ground pressure forces, the vertical loading and, overall, the running biomechanics.

DETAILED DESCRIPTION:
The analysis of the effects that listening to music may exert during exercise has been the topic of a number of scientific articles. Overall, these studies documented how music influences performance and they generally observed positive effects. The majority of the investigations were carried out in the aerobic/endurance domain where music was found to enhance running performance and is also likely to accelerate heart rate recovery after strenuous exercise, albeit not all the authors agree on this point. It has been also reported that loud music not only enhances optimal exercising, but also interacts with music tempo to yield significant additional performance benefits.

Despite such interesting findings, the focus of these investigations was restricted to characterize the physiological responses that individuals exhibit when listening to music during physical activity, mainly running. Thus, the studies ended up with positive results, that is, increased performance, or failed in showing any effect.

Beside the above reported positive effects of music some potentially negative effects should be considered. First, regardless of whether running is included or not in the experimental condition, exposure to high levels of noise/sound even for short periods of time can be damaging for the auditory system, possibly resulting in hearing loss or impairment. This topic has been scrutinized by a number of studies, with a specific attention to adolescent populations who are exposed to high risk of hearing problems due to the massive usage of listening devices. Although this is a crucial issue, such source of hazard can be adequately controlled for by firmly sticking to the guidelines on the recommended exposure limits (REL), which is recommended by the National Institute for Occupational Safety and Health (NIOSH). The REL has been set at 85 decibels (dB) for a maximum of 8 hours. Increasing the volume by rate of 3 dB increases the risk exponentially. For instance, a noise corresponding to an intensity of 88 dB should not exceed an exposure of 4 hours, then 91 dB 2 hours, 94 dB 1 hour, 97 dB 30 minutes, 100 dB 15 minutes, 103 dB 7.5 minutes, 106 dB 3.7 minutes and so on, up to 140 dB, which must not be provided at all.

Surprisingly, to date and to our knowledge, the influence that listening to music with portable devices and earphones may exert on the amount of vertical force upon impact loading during running has not been investigated yet.

Unlike the considerable number of previous works which were focused on the physiological and psychological responses to music during exercise, no references that attempted to address the biomechanical consequences of music listening on impact loading and jogging/running mechanics could be traced in the literature. Therefore, our main goal is to fill this gap in the existing literature.

Considering the universal widespread and popularity of running and that approximately 47 million Americans participated in running activities in the last decade, the findings generated by this research would be highly relevant to the broad field of sports medicine and exercise science.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age 18-35 years
* Level of fitness: Moderate level (ACTIVE) according to the classification of the American College of Sports Medicine depicting "Moderate" as either of the following 3 criteria:

  * 3 or more days of vigorous activity of at least 20 minutes per day OR
  * 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day OR
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 metabolic equivalents (METs) per week.
* able to run on a treadmill safely and without bilateral or unilateral support.

Exclusion Criteria:

* Past or present diseases of the auditory and vestibular system (as assessed by otolaryngological and audiometric examinations).
* Traumatology/orthopedic conditions that contraindicate treadmill training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Average ground pressure force | It will be assessed for each participant and for each arm of the study during the three 2-minute runs on the treadmill through study completion, an average of 1 year.
  This outcome expresses the mean amount of impact recorded by the force plates embedded in the treadmill.

SECONDARY OUTCOMES:
Peak ground pressure force | It will be assessed for each participant and for each arm of the study during the three 2-minute runs on the treadmill through study completion, an average of 1 year.
  This outcome expresses the highest amount of impact recorded by the force plates embedded in the treadmill.
Average vertical loading rate | It will be assessed for each participant and for each arm of the study during the three 2-minute runs on the treadmill through study completion, an average of 1 year.
  This outcome expresses the vertical oscillation of the center of mass and is considered highly linked to the risk of injury.
Stride length | It will be assessed for each participant and for each arm of the study during the three 2-minute runs on the treadmill through study completion, an average of 1 year.
  The stride length is the distance between two successive placements of the same foot.
Stride time | It will be assessed for each participant and for each arm of the study during the three 2-minute runs on the treadmill through study completion, an average of 1 year.
  It is the time elapsed between the first contact of two consecutive footsteps of the same foot and is expressed in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Manca Andrea, PhD, Principal Investigator — University of Sassari, Department of Biomedical Sciences; Franca Deriu, PhD, Study Director — University of Sassari, Department of Biomedical Sciences; Lucia Cugusi, PhD, Principal Investigator — University of Cagliari, Department of Medical Sciences and Public Health; Pomidori Luca, PhD, Principal Investigator — Esercizio Vita Medical Fitness; Felisatti Michele, PhD, Principal Investigator — Esercizio Vita Medical Fitness
Locations (2):
- Italy (2):
  - Department of Biomedical Sciences- University of Sassari, Sassari, Sassari (SS)
  - University of Sassari, Sassari

REFERENCES:
- [Background] Manca A, Cugusi L, Pomidori L, Felisatti M, Altavilla G, Zocca E, Zocca M, Bussu F, Dvir Z, Deriu F. Listening to music while running alters ground reaction forces: a study of acute exposure to varying speed and loudness levels in young women and men. Eur J Appl Physiol. 2020 Jun;120(6):1391-1401. doi: 10.1007/s00421-020-04371-z. Epub 2020 Apr 10. PMID 32277258
- [Background] Manca A, Cugusi L, Behm D, Dvir Z, Ferber R, Deriu F. More on "listening to music while running alters ground reaction forces": why women and men pound the ground differently? Eur J Appl Physiol. 2021 Jan;121(1):351-352. doi: 10.1007/s00421-020-04517-z. Epub 2020 Sep 30. No abstract available. PMID 32997258
- See also: NLM Pubmed — https://pubmed.ncbi.nlm.nih.gov/32277258/